CLINICAL TRIAL: NCT01332110
Title: Treatment for Patellofemoral Pain Syndrome Using Knee Abduction Moment-Reducing Footwear
Brief Title: Treatment for Patellofemoral Pain Syndrome Using Footwear
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ryan Lewinson, Ryan T. Lewinson, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23731
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Footwear; Motion Analysis; Running Injury
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Knee abduction moment-reducing footwear (Experimental): Footwear that is known to decrease knee abduction moments of force in healthy subjects. May include orthotics, or footwear that allows relative movement between the heel section of the outsole and rest of the shoe.
  Interventions: Device: Knee abduction moment-reducing footwear
- Control footwear (Placebo Comparator): Standard, off-the-shelf running shoes with no mechanical modifications.
  Interventions: Device: Knee abduction moment-reducing footwear

INTERVENTIONS:
Device: Knee abduction moment-reducing footwear — Patients in each study group will be asked to run using their assigned footwear at least 3 times per week (minimum 15 km per week) for six weeks. Each patient will document their perceived knee pain each week throughout the six week intervention.

SUMMARY:
Patellofemoral pain syndrome (PFPS) is the most common running injury and is believed to be associated with higher than normal knee joint loading. Footwear has been developed that may decrease these knee loads in healthy subjects, but their effects on patients with PFPS are unknown. In this study, we aim to test the effects of such footwear on patients with PFPS. We hypothesize that patients who receive the footwear intervention will show a decrease in knee joint loading, and consequently will show improvements in subjective levels of perceived knee pain over a period of six weeks compared to a control condition.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 18 and 45 years of age.
* Have been diagnosed with patellofemoral pain syndrome (PFPS) by a physician.
* Have nontraumatic unilateral and/or bilateral peripatellar or retropatellar knee pain.
* Patellofemoral knee pain with and/or after activity.
* Inactivity patellofemoral pain and/or stiffness, especially with sitting with knees held in flexed posture.
* Peripatellar tenderness ± mild inferior patellar pole tenderness.
* Run at least 15km per week.
* Are heel-toe runners (as opposed to forefoot strikers).

Exclusion Criteria:

* Are currently, or have previously, participated in any other forms of treatment for their knee pain.
* Significant articular or periarticular effusion or bursitis.
* Significant joint line tenderness.
* Intra-articular ligamentous instability.
* Patellar apprehension.
* Have undergone any form of knee surgery or arthroscopy.
* Have any other neuromuscular, musculoskeletal or cardiovascular conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Knee joint internal abduction moments of force during running at 4m/s | First day of joining the study
  Motion analysis trials will be conducted on each subject with both the control and intervention footwear. Inverse dynamics calculations will reveal the internal joint loading for each subject. Knee joint moments will be compared within subjects for each footwear condition.

SECONDARY OUTCOMES:
Change in subjective levels of perceived knee pain over six weeks | Upon initial recruitment to the study, and once per week for six weeks thereafter
  Pain levels will be recorded by 100mm visual analog scale during weeks 1, 2, 3, 4, 5 and 6 of the study to monitor the efficacy of the intervention. Final change in pain will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Darren J. Stefanyshyn, Ph.D. P.Eng., Principal Investigator — University of Calgary; Ryan T. Lewinson, B.Sc., Principal Investigator — University of Calgary; Jay T. Worobets, Ph.D., Principal Investigator — University of Calgary; J. Preston Wiley, M.D., M.P.E., Principal Investigator — University of Calgary
Locations (1):
- Human Performance Laboratory, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Lewinson RT, Wiley JP, Humble RN, Worobets JT, Stefanyshyn DJ. Altering Knee Abduction Angular Impulse Using Wedged Insoles for Treatment of Patellofemoral Pain in Runners: A Six-Week Randomized Controlled Trial. PLoS One. 2015 Jul 31;10(7):e0134461. doi: 10.1371/journal.pone.0134461. eCollection 2015. PMID 26230399